CLINICAL TRIAL: NCT00899912
Title: Investigating Markers of Radiation Outcome in Patients With Intermediate-Risk Prostate Cancer Using DNA Microarray Analysis: An RTOG Pilot Study
Brief Title: Changes in DNA After Radiation Therapy in Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RTOG-0612; CDR0000490025; NCI-2009-00734 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Microarray Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen tissue cores of prostatic biopsy specimens
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: microarray analysis
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Collecting and storing samples of tissue from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA after radiation therapy and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at changes in DNA after radiation therapy in patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Demonstrate the feasibility of acquiring specimens, both frozen and paraffin-embedded, to yield RNA of adequate quality to perform DNA microarray studies on markers of radiotherapy outcome in patients with intermediate-risk prostate cancer.

Secondary

* Compare the gene expression results from frozen tissue and paraffin-embedded tissue to see the correlation between the 2 methods in patients treated on the brachytherapy alone arm of protocol RTOG-0232.
* Find genes that are expressed differentially before and after radiation therapy in patients treated on the brachytherapy plus external-beam radiation therapy arm of protocol RTOG-0232.
* Find gene expression patterns in patients treated on either arm of protocol RTOG-0232 who have significant associations with biochemically as well as clinically apparent local and distant failure.

OUTLINE: This is a multicenter, pilot study.

Frozen and paraffin-embedded tissue samples are studied for biomarker/laboratory analysis. DNA microarray analysis is performed on the samples to assess markers of radiotherapy outcome.

PROJECTED ACCRUAL: A total of 156 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally confined adenocarcinoma of the prostate
* Zubrod performance 0-1
* Clinical stages T1c - T2b, N0, M0
* Combined Gleason score 7 if prostate specific antigen (PSA) < 10, combined Gleason score < 7 if PSA 10 - 20; PSA must be ≤ 20 ng/mL, before hormone therapy, if given, and a prostate volume by transrectal ultrasound (TRUS) ≤ 60 cc.
* American Urological Association (AUA) score ≤ 15 (alpha blockers are allowed).
* Age ≥ 18 years old and must sign a study-specific informed consent form

Exclusion Criteria:

* No clinically or pathologically involved lymph nodes
* No distant metastases or significant obstructive symptoms
* No prior chemotherapy, pelvic radiation, transurethral prostatectomy (TURP), cryosurgery, TUNA, transurethral microwave thermotherapy (TUMT) or radical surgery for carcinoma of the prostate is allowed.
* No previous hormonal therapy beginning < 2 months or > 6 months prior to registration is allowed.
* No previous or concurrent cancers other than basal, in situ, or squamous cell skin cancers unless the patient is disease free for ≥ 5 years.
* No hip prosthesis or major medical or psychiatric illnesses are allowed. prior to study entry.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intermediate risk prostate cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of frozen and paraffin-embedded specimens that yield adequate RNA for tumor tissue microarray analysis | Specimens collected at the time of brachytherapy

SECONDARY OUTCOMES:
Comparison of gene expression patterns between frozen and paraffin-embedded tissue in patients treated on the brachytherapy alone arm of protocol RTOG-0232 | After microarray analysis of tissue and primary endpoint analysis of RTOG 0232
Comparison of genes to determine which are expressed differentially before and after radiotherapy in patients treated on the brachytherapy plus external-beam radiation therapy arm of protocol RTOG-0232 | After microarray analysis of tissue and primary endpoint analysis of RTOG 0232
Gene expression patterns in patients treated on either arm of protocol RTOG-0232 who have significant associations with biochemically as well as clinically apparent local and distant failure | After microarray analysis of tissue and primary endpoint analysis of RTOG 0232

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Chakravarti, MD, Study Chair — Ohio State University
Locations (10):
- United States (10):
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania